CLINICAL TRIAL: NCT03818529
Title: US Cohort Study of Previously Untreated Patients (PUPs) With Congenital Hemophilia
Brief Title: ATHN 8: Previously Untreated Patients (PUPs) Matter Study
Status: Completed | Type: Observational
Sponsor: American Thrombosis and Hemostasis Network (Network)
Collaborators: CSL Behring (Industry); Octapharma (Industry); Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: ATHN 8
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Hemophilia; Hemophilia A; Hemophilia B; Hemophilia A With Inhibitor; Hemophilia B With Inhibitor; Haemophilia B Without Inhibitor; Haemophilia A Without Inhibitor; Haemophilia
Keywords: Hemophilia; Previously Untreated Patients (PUPs); Clotting Factor Replacement Products; Haemophilia
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center cohort study of approximately 250 previously untreated patients (PUPs) with congenital moderate to severe hemophilia A or B in a network of up to 50 US Hemophilia Treatment Centers (HTCs). Participants will be followed as they receive their first 50 exposure days (ED) to clotting factor replacement product, both prospectively and retrospectively. The data collected on evolving treatment practices will define the incidence and risk factors for inhibitor development during the high risk period of first 50 ED and improve the outcomes of this vulnerable population.

DETAILED DESCRIPTION:
This multi-center, longitudinal, observational, prospective and retrospective study of previously untreated patients (PUPs) with moderate to severe hemophilia A or B during the initial 50 exposure days (ED) to clotting factor replacement product or until the development of a confirmed inhibitor. The Primary Investigators have designed the study to utilize the American Thrombosis and Hemostasis Network (ATHN) electronic infrastructure to leverage existing data and enable the collection of more in-depth clinical and laboratory data on PUPs. The study aligns with the National Hemophilia Foundation Medical and Scientific Advisory Council (MASAC) recently issued Recommendation #243 which includes: "Regardless of which option is chosen, all PUPs should be enrolled in the ATHN data collection system or a clinical trial to assess outcomes." Co-enrollment in the ATHNdataset by participants is required. The total study duration is planned for 6 years.

The primary objective is to determine the percentage of patients with confirmed inhibitors within the first 50 ED. Confirmed inhibitors are defined as two consecutive positive inhibitor titers (per CDC laboratory criteria; >0.5 Nijmegen Bethesda Units for hemophilia A and >0.3 Nijmegen Bethesda Units for hemophilia B) on different blood samples which result in change in treatment recommendations.

Please note - the treatment regimen will be at the discretion of the participants' hemophilia caregivers. No treatment products are being provided by the study nor will the participants be paid. However, inhibitor titer testing will be provided at no cost to participants by the Centers for Disease Control and Prevention (CDC).

All study procedures and follow-up will be timed to coincide with scheduled hemophilia care whenever possible. Ad hoc, quarterly follow-up, annual and final visits are for participants who have not met study endpoints (50 ED or inhibitor development) prior to enrollment.

Data collected will include eligibility, demographics, medical history (co-morbidities, surgery/procedures, immunizations and allergies), hemophilia history (severity, genotype and family history), birth history, inhibitor testing results, detailed treatment product(s) usage, bleeding events, bleeding disorder related medical visits during the study, and EUHASS adverse events.

Sub-studies

A number of sub-studies are planned with pharmaceutical sponsors to collect information from patients about their specific product use. Participation in these product specific sub-studies is optional and sub-study visits will be planned to coincide with HTC visits. The sub-study will collect information from patients about their perception and use of treatment products, physical activity levels and other general health questions. This data will be collected via questionnaire.

Data Collection System

All data collected will be entered into electronic case report forms (eCRFs) within the secure ATHN System by HTC site personnel. All participating study sites will have in place a current, executed Data Use and Business Associate Agreement (DUBAA) with ATHN.

ELIGIBILITY:
Inclusion Criteria:

* Congenital hemophilia A; FVIII </=5% or congenital hemophilia B; FIX </=5%;
* Birth date on or after January 1, 2010;
* Care established at one of the participating HTCs;
* Co-enrollment in the ATHNdataset; and
* Parent or authorized guardian can provide informed consent

Exclusion Criteria:

* Patients who are referred to the HTC with no record of bleed and factor utilization data

Ages: 0 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will enroll a cohort of 250 participants born with hemophilia on or after January 1, 2010 who meet the eligibility criteria and are receiving care from one of the participating HTCs.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Determine percentage of patients with confirmed inhibitors | 6 years
  Participants will be followed to assess inhibitor development (per CDC laboratory criteria; >0.5 Nijmegen Bethesda Units for hemophilia A and >0.3 Nijmegen Bethesda Units for hemophilia B) within 50 exposure days. Blood specimens will be submitted to the CDC for inhibitor testing at various time points outlined in the protocol.

SECONDARY OUTCOMES:
Determine risk factors including genetic variants associated with inhibitor development in PUPs | 6 years
  The study will provide a systematic approach to data collection by using the ATHN System to provide database infrastructure and data collection methods to evaluate determinants of inhibitor formation.
Determine percentage of eligible participants enrolled at each site | 6 years
  Sites will report number of eligible participants and number of participants enrolled to determine the percentage of enrollment.
Determine mean age of diagnosis and first exposure to factor treatment product | 6 years
  Sites will document the date of diagnosis and the date of first exposure to clotting factor treatment product.
Determine the number of exposure days prior to inhibitor development | 6 years
  Sites and participants will work together to provide detailed records of exposure days to clotting factor replacement products. The CDC will act as the central laboratory for the study and provide inhibitor testing.
Report bleeding complications that occur within the first 50 ED | 6 years
  The documentation of bleeding events in the study records will be based on the review of bleeding and infusion records provided by the participant or the from medical chart review during the first 50 exposure days to clotting factor replacement product.
Summarize factor replacement dosing regimen prescribed to this study population within the first 50 ED | 6 years
  A summary of the prescribed clotting factor replacement regimen will provide data on evolving treatment practices, including specific clotting factor replacement and non-factor products.
Report on the number of transient inhibitor, e.g., those which resolve without change in therapy | 6 years
  The CDC is acting as the central laboratory for inhibitor testing. The CDC will report results to the participating HTC. If a blood specimen from a participant has an elevated result; potentially indicating the development of an inhibitor, a new blood specimen from the participant will be tested within 10 days of the first elevated result to determine if an inhibitor has developed. A transient inhibitor is defined as a positive inhibitor which is not confirmed on a consecutive repeat testing. Inhibitor testing results on all participants will be documented and reported by the HTC.
Report on targeted post-approval safety data for events related to clotting factor replacement products used by prospectively enroll participants | 6 years
  Documentation of adverse events experienced by prospectively enrolled participants during the study period of first 50 exposure days to clotting factor replacement product will be reported. The types of adverse events to be reported are limited to Serious Adverse Events as defined by the European Union Haemophilia Safety Surveillance System (EUHASS).
Sub-study modules will be developed to evaluate and report on cohorts of study participants who initiated treatment with a specific product | 6 years
  Measure the number of participants who initiate treatment with a specific treatment product

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Carpenter, MD, MS, Principal Investigator — Children's Mercy Hospital Kansas City; Courtney Thornburg, MD, MS, Principal Investigator — University of California San Diego, Rady Children's Hospital San Diego; Marijke van den Berg, MD, PhD, Principal Investigator — Versiti Blood Health
Locations (27):
- United States (27):
  - Arizona Hemophilia and Thrombosis Center at Phoenix Children's Hospital, Phoenix, Arizona
  - Valley Children's Hospital, Madera, California
  - Rady Children's Hospital San Diego, San Diego, California
  - UCSF Pediatric Hemophilia Treatment Center at Mission Bay, San Francisco, California
  - University of Colorado Denver Hemophilia and Thrombosis Center, Aurora, Colorado
  - Connecticut Bleeding and Clotting Disorders Center, Farmington, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta/Emory, Atlanta, Georgia
  - Augusta University Hemophilia Treatment Center, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center (IHTC), Indianapolis, Indiana
  - Kansas City Regional Hemophilia Center, Kansas City, Kansas
  - Maine Hemophilia and Thrombosis Center, Scarborough, Maine
  - Boston Hemophilia Center at Children's Hospital of Boston, Boston, Massachusetts
  - University of Michigan Hemophilia and Coagulation Disorders, Ann Arbor, Michigan
  - Mayo Comprehensive Hemophilia Center, Rochester, Minnesota
  - Cincinnati Children's Hospital Medical Center, Hemophilia & Thrombosis Center, Cincinnati, Ohio
  - UHHS Cleveland, Cleveland, Ohio
  - Northwest Ohio Hemophilia Treatment Center at the Toledo Hospital, Toledo, Ohio
  - Oklahoma Center for Bleeding and Clotting Disorders, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Utah Center for Bleeding & Clotting Disorders at Primary Children's Hospital, Salt Lake City, Utah
  - Hemophilia Outreach Center, Green Bay, Wisconsin
  - Blood Center of Wisconsin, Milwaukee, Wisconsin